CLINICAL TRIAL: NCT01931865
Title: IncobotulinumtoxinA for Treatment of Focal Cancer Pain After Surgery and/or Radiation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lost the recruiting source- no recruitment for the past 18months, PI moving
Sponsor: Yale University (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205010328
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: cancer pain, radiation therapy, surgery, incobotulinum toxin
MeSH Terms: conditions — Pain; Cancer Pain | interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IncobotulinumtoxinA (Experimental): The total dose will depend on the extent of the area involved by pain. The injections will be carried out through a 1cc syringe using a ½ to 1 inch needle intramuscularly or subcutaneously (or both). The ttoal dose will not exceed 100 units.
  Interventions: Drug: IncobotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Subject will receive Xeomin, injected into the area of reported focal pain associated with prior cancer treatment. The total dose will depend on the extent of the area involved by pain. botulinum toxin which is marketed under the trade name of Xeomin. Xeomin is approved by FDA for certain conditions.
  Other Names: Xeomin

SUMMARY:
The purpose of this research study is to investigate the safety and effectiveness of botulinum toxin A (Xeomin) ® injections in patients who suffer from focal pain in areas of radiation and/or surgery as a result of cancer treatment. Our hypothesis is that injection of incobotulinum toxin A into an area of local pain, at or around the area of a post-surgical/post radiation scar, relieves the focal cancer pain.

DETAILED DESCRIPTION:
Please contact the PI for more detailed information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18- 80 years, both sexes, all races and ethnic groups.
* Diagnosis of post- surgical/post - radiation cancer pain.
* Focal pain duration longer than 3 months
* Pain of moderate to severe intensity ( mean VAS over the previous week >4 )
* Subjects who are able to read, speak, and understand English.

Exclusion Criteria:

* Existing significant acute medical condition (i.e. cardiovascular, endocrine, hematologic, neoplastic, infectious, or autoimmune disorders).
* Pregnancy or planned pregnancy (determined by urine pregnancy test). Women of childbearing age should use a reliable mode of contraception during the study period (abstinence, etc).
* Active breast feeding.
* Enrollment in any clinical trial (currently or within the past 3 months) in which treatments are imposed by a protocol.
* Any subject for whom botulinum toxin treatment would be contraindicated; known allergy or sensitivity to medication.
* Subjects who are younger than 18 years of age.
* Neuromuscular-junction disorders.
* Axis I diagnosis determined by a neurologist or psychiatrist.
* Use of anesthetic medications within two weeks or corticosteroid injections within 4 weeks of enrollment.
* Received botulinum toxin injections in the past 4 months.
* Patients taking high doses of aminoglycosides or other drugs affecting the function of neuromuscular junction ( anticholinergic, muscle relaxants)
* Patients who have unstable pain in/at sites other than areas of planned injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Jabbari, MD, Principal Investigator — Yale University
Locations (1):
- Yale Physician Building, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IncobotulinumtoxinA: The total dose will depend on the extent of the area involved by pain. The injections will be carried out through a 1cc syringe using a ½ to 1 inch needle intramuscularly or subcutaneously (or both). The number of injections will not exceed 5 sites.
  IncobotulinumtoxinA: Subject will receive Xeomin, injected into the area of reported focal pain associated with prior cancer treatment. The total dose will depend on the extent of the area involved by pain. botulinum toxin which is marketed under the trade name of Xeomin. Xeomin is approved by FDA for certain conditions.
Period: Overall Study
Arm/Group | IncobotulinumtoxinA
Started | 12
Completed | 8
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | IncobotulinumtoxinA
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Significant Reduction in Pain
Description: visual analogue scale (VAS), a line which represents the level of pain in 10cms and you will show where your pain is on this line (0 no pain, 10 worst pain). A significant reduction is 2 grades on the scale.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA
Number analyzed (Participants) | 8
participants | 8

2. Secondary Outcome: Patients Who Show Improvement in American Pain Association Questionnaire
Description: This quality of life scale consists of 10 questions regarding how pain affects your quality of life.
Time Frame: 12 weeks
Population: Advanced cancer patients
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA
Number analyzed (Participants) | 8
participants | 3

3. Other Pre Specified Outcome: Patients Improved in Patient Global Impression of Change (PGIC) Scale
Description: The Patient Global Impression of Change questionaire asks patient level of satisfaction with current treatment (from very unsatisfactory to very satisfactory).
Time Frame: 12 weeks
Population: Advanced cancer patients
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA
Number analyzed (Participants) | 8
participants | 7

ADVERSE EVENTS:
Time Frame: 3 months- Advised to call the adverse effect immediately
Arm/Group | IncobotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Open study, small number of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No